CLINICAL TRIAL: NCT01914029
Title: Immunological Mechanisms of Allergy Immunotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 0032-13-RMB CTIL
Record Dates: First submitted 2013-06-06; First posted 2013-08-01 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Allergy Desensitization

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the study is to add to the knowledge of mechanisms of immune health. Parameters of the immune system will be followed over time in volunteers allergic to dust mites and bee sting after receiving immunization therapy. This information will be compared to healthy volunteers without allergy. We aim to bring new understanding of immune processes by this comparison.

DETAILED DESCRIPTION:
The process of immunization as a treatment for allergic disease brings about changes that are not all well understood and the understanding about them is developing constantly. In our study we plan to check a large number of immunological parameters to broaden the scope of knowledge of evaluating individuals for immune health across multiple sub fields of medicine and for advancing a basic understanding of immune cell signaling.

The study will involve 70 participants between ages 18-45 of both sexes. Persons enrolled to the study will have been diagnosed with allergic rhinitis caused by dust mite or persons who developed a systemic reaction following bee sting who are candidates to be treated by immunization.

After verification of diagnosis of allergic condition and decision to start immunizations, blood samples will be drawn from participants before immunization weekly for 24 weeks. Blood samples will be analyzed in order to identify immune cell subset differences that change in response to allergy immunotherapy. Comparisons will be made of baseline and stimulation-induced status of protein phosphorylation individuals over the time-series course in which they receive allergy immunotherapy to pinpoint molecular mechanisms underlying desensitization. Evaluations will be made of cellular mechanisms of allergy immunotherapy by comparing over time and between groups, through serum cytokine profiling and blood gene expression of individuals undergoing allergy immunotherapy shots.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of allergic rhinitis and evidence of specific immunoglobulin E antibodies to house dust mite.

Or A history of a bee sting event that resulted in a systemic allergic reaction with evidence of bee venom-specific immunoglobulin E by skin testing 18-45 years, inclusive at time of initial enrollment General good health and ambulatory at time of enrollment Willing and able to sign Informed Consent Available for follow-up for the planned duration of the study Acceptable medical history by screening evaluation and brief clinical assessment

-

Exclusion Criteria:

Allergy to multiple allergens Active systemic or serious concurrent illness, including febrile illness on the day of blood withdrawal History of immunodeficiency Known or suspected impairment of immunologic function, including, but not limited to clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease, blood pressure >150/95 at screening, or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.

Chronic Hepatitis B or C. Recent or current use of immunosuppressive medication, including glucocorticoids (corticosteroid nasal sprays are permissible).

Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).

Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.

History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin, Plavix, Aggrenox. May be acceptable after review by investigator.

Receipt of blood or blood products within the past 6 months Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol History of Guillain-Barré Syndrome

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 10 volunteers will be enrolled in each group. The study will include seven treatment groups and one control, total number of participants is 80
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Immunological changes within allergic desensitization treatment | 1. Immunological changes from baseline to 4 months
  1. Phenotype changes in time of immune cell subsets count, and relative abundance.
  2. Compare the baseline and stimulation-induced status of protein phosphorylation individuals over the time-series course in which they receive allergy immunotherapy and pinpoint molecular mechanisms underlying desensitization.
  3. Evaluate cellular mechanisms of allergy immunotherapy by comparing over time and between groups, through serum cytokine profiling and blood gene expression of individuals undergoing allergy immunotherapy shots.

SECONDARY OUTCOMES:
Allergen Immunotherapy | participants will be followed weekly for 4 months and once a month afterwards for a year
  Compare the baseline and stimulation-induced status of protein phosphorylation individuals over the time-series course in which they receive allergy immunotherapy and pinpoint molecular mechanisms underlying desensitization.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Shahar, Dr., Principal Investigator — Rambam Health Care Campus
Locations (1):
- Immunology Clinic Rambam Medical Center, Haifa, Israel